CLINICAL TRIAL: NCT07176702
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination With Trastuzumab and Chemotherapy for the First-Line Treatment of HER2-Positive Pancreatic Ductal Adenocarcinoma
Brief Title: A Phase II Clinical Study of HLX22 in Combination With Trastuzumab and Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Liang Liu, Professor & Chief Physician, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX22-IIT-PDAC201
Record Dates: First submitted 2025-08-26; First posted 2025-09-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic PDAC; HER2-positive Status
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia | interventions — Trastuzumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX22 in Combination with Trastuzumab and Chemotherapy (Experimental)
  Interventions: Drug: HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination with Trastuzumab and Chemotherapy

INTERVENTIONS:
Drug: HLX22 (Recombinant Humanized Anti-HER2 Monoclonal Antibody Injection) in Combination with Trastuzumab and Chemotherapy — Drugs: HLX22 (15 mg/kg IV) + trastuzumab (8 mg/kg loading dose → 6 mg/kg maintenance) + nab-paclitaxel (125 mg/m² IV) + gemcitabine (1000 mg/m² IV).
  Administration: Administered every 3 weeks until disease progression, unacceptable toxicity, or withdrawal.

SUMMARY:
Pancreatic cancer is an extremely high-mortality malignancy. The chemotherapy regimen of gemcitabine combined with nab-paclitaxel (GEM-NABP) serves as one of the first-line standard therapies for metastatic pancreatic cancer. Given that traditional dual HER2 blockade (pertuzumab + trastuzumab) has demonstrated preliminary efficacy in HER2-expressing solid tumors, the novel clinical strategy of dual HER2 blockade (HLX22 + trastuzumab) combined with GEM-NAP offers the potential to improve outcomes for patients with HER2-positive pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary Participation Willingly participate in the clinical study; fully comprehend the study details and sign the Informed Consent Form (ICF); commit to and demonstrate capacity to complete all trial procedures.
* Age and Gender Any gender; age ≥18 and ≤75 years at the time of ICF signing.
* Diagnosis Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma (PDAC).
* Prior Therapy *No prior systemic antitumor therapy for metastatic PDAC.

  *Exception: Patients who received one cycle of chemotherapy (nab-paclitaxel + gemcitabine) as initial treatment for newly diagnosed PDAC may enroll.

  *Prior neoadjuvant/adjuvant therapy is permitted if completed >6 months before enrollment, and treatment-related adverse events (AEs) have recovered to NCI-CTCAE ≤ Grade 1 (alopecia excluded).
* Measurable Disease At least one measurable lesion per RECIST v1.1, assessed by the investigator. Target lesions must not be exclusively bone metastases.
* HER2 Status *HER2-positive defined by ASCO/CAP gastric cancer HER2 testing guidelines: IHC 3+ (primary or metastatic lesion), or IHC 2+ with ISH/FISH-positive confirmation.

  *Note: ≤15 patients with IHC 2+/FISH-positive status may enroll.
* Performance Status ECOG performance status 0 or 1 within 7 days prior to first dose.
* Life Expectancy Expected survival ≥3 months.
* Hepatitis B *HBsAg-negative and HBcAb-negative. *If HBsAg-positive or HBcAb-positive, HBV-DNA must be <2500 copies/mL or 500 IU/mL (or within institutional normal range).
* Hepatitis C *HCV antibody-negative.

  * If HCV antibody-positive, HCV-RNA must be negative.
  * Exclusion: Co-infection of HBV and HCV (HBsAg/HBcAb-positive and HCV antibody-positive).
* HIV Status HIV antibody-negative.
* Organ Function

Adequate organ function within 14 days before first dose (without transfusion, albumin, thrombopoietin, or CSF support):

*Hematology: Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L Platelets ≥100 × 10⁹/L Hemoglobin ≥90 g/L

*Liver: Total bilirubin ≤1.5 × ULN AST/ALT ≤2.5 × ULN (≤5 × ULN if liver metastases present) Alkaline phosphatase ≤5.0 × ULN Albumin ≥25 g/L

*Renal: Creatinine clearance ≥50 mL/min (Cockcroft-Gault formula)

*Coagulation: INR ≤1.5 × ULN APTT ≤1.5 × ULN PT ≤1.5 × ULN

* Contraception

  * Females of childbearing potential: Negative serum pregnancy test within 7 days before first dose.
  * All participants: Use of ≥1 medically approved contraceptive method (e.g., IUD, oral contraceptives, barrier devices) during treatment and for ≥7 months after last dose.

Exclusion Criteria:

* Other Malignancies

History of other malignancies within 2 years prior to first dose, except:

Curatively treated localized tumors (e.g., basal cell carcinoma, squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of prostate/cervix/breast/thyroid).

* Prior Anthracycline Exposure

Cumulative doxorubicin dose > 360 mg/m² (or equivalent):

Equivalent agents: Epirubicin >720 mg/m², mitoxantrone >120 mg/m², idarubicin >90 mg/m², or liposomal doxorubicin >360 mg/m² doxorubicin-equivalent.

If multiple anthracyclines were used, the total cumulative dose must not exceed 360 mg/m² doxorubicin-equivalent.

* Prior HER2-Targeted Therapy Any previous HER2-targeted treatment (e.g., trastuzumab, pertuzumab).
* Active Gastrointestinal Bleeding

  ≥ Grade 2 toxicity per NCI-CTCAE v5.0.
* CNS Involvement Central nervous system (CNS) metastases and/or leptomeningeal metastases.
* Cardiovascular Events

History within 6 months prior to first dose:

Cerebrovascular accident, myocardial infarction, unstable angina, or poorly controlled arrhythmias.

QTc interval ≥450 ms (males) or ≥470 ms (females) (Fridericia formula).

* Cardiac Dysfunction NYHA Class III-IV heart failure or left ventricular ejection fraction (LVEF) < 55% by echocardiography.
* Pulmonary/Infectious Conditions Interstitial lung disease (current or history). Active infection requiring systemic therapy or active tuberculosis.
* Recent Live Vaccines Administration of live attenuated vaccines within 28 days prior to first dose (exception: inactivated influenza or COVID-19 vaccines).
* Major Surgery Within 28 days prior to first dose.
* Radiotherapy Curative radiotherapy within 28 days prior to first dose.
* Concurrent Clinical Trials Current participation in other interventional studies or use of investigational drugs/devices within 28 days prior to first dose.
* Hypersensitivity Known severe allergy to monoclonal antibodies or excipients of the study drugs.
* Substance Abuse History of illicit drug use or psychiatric medication abuse.
* Pregnancy/Lactation Pregnant or breastfeeding women.
* Other Exclusionary Factors

Any condition deemed by the investigator to:

Compromise patient safety or data integrity. Require concomitant treatment for severe comorbidities (including psychiatric disorders).

Exhibit critically abnormal laboratory values. Pose significant social/familial impediments to study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-03-05 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by investigators per RECIST v1.1. | up to 36 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 12 months
Overall Survival (OS) | up to 36 months
Disease Control Rate (DCR) | up to 36months
Duration of Response (DOR) | up to 36 months
Incidence of Adverse Events (AEs) | up to 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Drum Tower Hospital, Nanjing, Nanjing
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality